CLINICAL TRIAL: NCT04425772
Title: A Randomized,Double Blinded, Double Dummy, Parallel Controlled Clinical Trial for Azvudine in the Treatment of Novel Coronavirus Pneumonia (COVID-19）
Brief Title: A Clinical Trial for Azvudine in the Treatment of Novel Coronavirus Pneumonia (COVID-19）
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Genuine Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FNC-Hope4
Record Dates: First submitted 2020-05-09; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): FNC+Standard of Care
  Interventions: Drug: FNC+Standard of Care
- Control Group (Placebo Comparator): FNC dummy tablet+ Standard of Care
  Interventions: Drug: FNC dummy tablet+Standard of Care

INTERVENTIONS:
Drug: FNC+Standard of Care — FNC + Standard of Care according to the to the latest version of the National Health and Medical Commission Diagnostic criteria
  Other Names: Azvudine+SOC
  Arms: Experimental Group
Drug: FNC dummy tablet+Standard of Care — FNC dummy tablet+ Standard of Care according to the to the latest version of the National Health and Medical Commission Diagnostic criteria
  Other Names: Azvudin dummy tablet+SOC
  Arms: Control Group

SUMMARY:
To evaluate the efficacy and safety of azvudine in treatment of COVID-19

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years old, gender not limited;
2. Laboratory (RT-PCR) confirmed COVID-19;
3. the time from the first positive nucleic acid test to randomization does not exceed more than 4 days;
4. informed consent has been signed.

Exclusion Criteria:

1. known or suspected allergies to the components of azivudine tablets;
2. according to the latest version of the National Health and Medical Commission Diagnostic criteria of COVID-19, patients with severe novel coronavirus pneumonia was confirmed;
3. severe liver disease (TBIL>=2 times normal upper limit; ALTAST>=5 times normal upper limit);
4. subjects with severe renal insufficiency (glomerular filtration rate ≤60 mL/min/1.73 m2) or undergoing continuous renal replacement therapy, hemodialysis or peritoneal dialysis;
5. subjects with complication of malabsorption syndrome or any other condition affecting gastrointestinal absorption, requiring intravenous nutrition or not being able to take drugs orally;
6. subjectsis currently receiving anti-hiv treatment;
7. women who are breast-feeding during pregnancy or have a family plan during the trial period and within 6 months after the end of the trial;
8. participating in other clinical trials or using experimental drugs, except traditional Chinese medicine;
9. Other conditions that not appropriate to be enrolled into this study based on investigator's advise.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Estimated)
Dates: Start 2020-06-12 (Estimated); Primary Completion 2020-08-12 (Estimated); Study Completion 2020-08-12 (Estimated)

PRIMARY OUTCOMES:
Change (reduction) in viral load from baseline | On day 7 and 14
  (reduction) in viral load from baseline

SECONDARY OUTCOMES:
proportion of subjects change from mild or moderate type to severe type | up to 21 days
  proportion of subjects change from mild or moderate type to severe type
proportion of subjects change from severe type to critical type | up to 21 days
  proportion of subjects change from severe type to critical type
novel coronavirus nucleic acid conversion rate | up to 21 days
  novel coronavirus nucleic acid conversion rate
Novel coronavirus nucleic acid negative conversion time | up to 21 days
  Novel coronavirus nucleic acid negative conversion time
The time and proportion of improvement in pulmonary imaging | up to 21 days
  TIme(Days);Proportion(percent)
Time and proportion of temperature return to normal | up to 21 days
  TIme(Days);Proportion(percent)
time and rate of improvement of respiratory symptoms and signs (lung rhones, cough, sputum, sore throat, etc.) | up to 21 days
  TIme(Days);Proportion(percent)
time and rate of improvement of diarrhea, myalgia, fatigue and other symptoms | up to 21 days
  TIme(Days);Proportion(percent)
Changes of blood oxygen detection index | up to 21 days
  Changes of blood oxygen detection index
Frequency of requirement for supplemental oxygen or non-invasive ventilation | up to 21 days
  Frequency of requirement for supplemental oxygen or non-invasive ventilation
Frequency of adverse events | up to 21 days
  Frequency of adverse events